CLINICAL TRIAL: NCT06869252
Title: Autologous Adipose Cells Therapy
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CERM INC. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CERM 002
Record Dates: First submitted 2025-02-27; First posted 2025-03-11 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Hair Loss/Baldness; Wrinkle Appearance; Volume; Fine Lines; Skin Elasticity; Hair Thinning; Skin Pigmentation; Skin Texture
Keywords: Adipose Cells; Adipocytes
MeSH Terms: conditions — Alopecia; Pigmentation Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Autologous Adipose Cells Therapy (Experimental)
  Interventions: Biological: Autologous Adipose Cells Therapy

INTERVENTIONS:
Biological: Autologous Adipose Cells Therapy — Participants will receive Autologous Adipose Cells therapy treatment, and the safety and efficacy of the treatment will be monitored by the primary investigator up to 25 weeks.

SUMMARY:
Autologous Adipose Cell Therapy is a series of process designated to address the demerits of the traditional autologous fat grafting and dermal fillers, while enhancing the versatility and aesthetic outcomes. In this study, the goal is to evaluate the safety and efficacy of Autologous Adipose cell Therapy for skin rejuvenation and hair improvement in human application.

DETAILED DESCRIPTION:
Autologous fat grafting (AFG) and injection of dermal fillers are the most prevailing aesthetic procedures in the cosmetic field for skin rejuvenation and hair restoration. High degree of biocompatibility and biodegradability of dermal fillers contribute significantly to their effectiveness in skin rejuvenation and hair restoration; however, the results are typically not enduring. On the other hand, autologous fat grafting is increasingly recognized for its applications not only in skin rejuvenation, but also breast augmentation and the treatment of arthritis. Fat fillers are fully biocompatible to the recipient, due to the use of autologous cell, the effects generally persist longer than those achieved with dermal fillers. Nonetheless, unprocessed lipoaspirate collected through liposuction procedure has a heterogeneous composition, which potentially leads to uneven distribution of adipose tissu resulting in formation of lumps or nodules at the recipient's site. Volume retention following autologous fat grafting is not solely affected by the resorption rate of adipose cells, but also impacted by re-uptake rate of other components of lipoaspirate. Autologous Adipose Cell Therapy seeks to enhance the current autologous fat grafting by isolating early-stage adipose cells from lipoaspirate and optimizing the number of adipocytes cells within the fat filler through cell property of differentiation. The purpose of this study is to assess the safety, feasibility, and efficacy of Autologous Adipose Cell Therapy for skin rejuvenation and hair improvement in human subjects. The eligibility of participants who are interested in participating in this study will be determined based on the inclusion and exclusion criteria listed in the study protocol. The in-charge plastic surgeon will monitor and evaluate the treatment outcomes in participants over a six-months period after the administration of Autologous Adipose Cell Therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatients who express interest in skin rejuvenation, and/or who are experiencing skin conditions, such as winkles, fine lines, loss of skin elasticity, skin pigmentation, scarring.
2. Outpatients who are experiencing hair loss or hair thinning
3. Provision of signed and dated informed consent form
4. Clearly stated willingness to comply with all the procedures of the study and availability of the study
5. Female and Male aged between 21 to 80 years old 6 Medical clearance by family doctor

Exclusion Criteria:

1. Pregnancy or lactation
2. Known allergic reaction to components of cell culture media
3. Chronic disease , e.g. cardiovascular disease, diabetes, chronic kidney disease, seizures
4. Chronic infections, e.g. skin fungi infection, psoriasis
5. Chronic wound healing
6. Currently taking hormone therapy
7. History of cancers and active cancers
8. Viral infection, e.g. HIV, hepatitis B, influenza, coronaviruses.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Outcome Comparison Survey | The end of the study (Week 20 to 25)
  30 people will be randomly selected to rank the level of improvement by comparing the images captured at pro and post-treatment from Imaging assessment.
  Scale of Improvement:
  * No Improvement(0%)
  * Minimal Improvement(1% - 25%)
  * Moderate Improvement(26% - 50%)
  * Significant Improvement(51% - 75%)
  * Major Improvement(76% - 100%)
Participant Satisfaction Survey | From first post-treatment follow-up visit to the last follow-up visit at week 16 to week 25
  Participants will be requested to complete a list of questions related to their experience and satisfaction of autologous adipose cell therapy in each study visit for result evaluation.
  1-to-5 Scales:
  * 1 being "very poor" and 5 being "excellent"
  * 1 being "very dissatisfied" and 5 being "very satisfied"
Imaging Assessment | From first pre-treatment visit to the last follow-up visit at week 16 to week 25
  Digital images of the target site will be captured for each participant both prior to and following autologous adipose cell therapy for the purpose of outcome evaluation. The comparison of pre- and post-treatment images will be utilized in the "Outcome Comparison Survey" and the "Visit Evaluation Report" to assess the degree of improvement, based on the established assessment parameters for Autologous Adipose Cell Therapy treatment.
Case Report Form | The report will be completed at the end of the study (Week 20 to 25), but highlights would be recorded in this document during every visit.
  A comprehensive medical document will be prepared by the responsible plastic surgeon which outlines the key details of each stage of the treatment process and aspects based on each participant's case. This document will include a thorough description of the patient's presenting medical conditions, the surgical procedures performed, post-treatment progress, any adverse events that occurred, and the final outcomes.
Visit Evaluation Report | From first post-treatment follow-up visit to the last follow-up visit at week 16 to week 25
  During each post-treatment visit, the responsible plastic surgeon will assess the treatment outcomes and evaluate the degree of improvement by comparing the pre-treatment image with the current post-treatment image.
  Scale of Improvement:
  * No Improvement(0%)
  * Minimal Improvement(1% - 25%)
  * Moderate Improvement(26% - 50%)
  * Significant Improvement(51% - 75%)
  * Major Improvement(76% - 100%)
  Assessment Parameters:
  Skin:
  * Radiance
  * Texture
  * Firmness
  * Wrinkles & Fine Lines
  * Spot Hyperpigmentation
  * Tone
  * Redness & Inflammation
  * Pore Size
  Hair:
  * Density
  * Thickness
  * Visual Appearance
  * Texture (Smoothness & Frizz Control)
  * Shine
  * Scalp Health

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Abdollah M. Malekzadeh, MD, MD, Principal Investigator — The Centre for Cosmetic Surgery & Medicine; Dr. Arun Kumar, PhD, Study Director — CERM INC.
Locations (2):
- United States (2):
  - The Centre for Cosmetic Surgery & Medicine, Newark, Lewes, Delaware
  - The Centre for Cosmetic Surgery & Medicine, Newark, Delaware

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bellini E, Grieco MP, Raposio E. The science behind autologous fat grafting. Ann Med Surg (Lond). 2017 Nov 10;24:65-73. doi: 10.1016/j.amsu.2017.11.001. eCollection 2017 Dec. PMID 29188051
- [Background] Sutcliffe H, Rawlinson PS, Thakker B, Neary R, Mallick N. Factitious proteinuria: diagnosis and protein identification by use of isoelectric focusing. Clin Chem. 1988 Aug;34(8):1653-5. PMID 3402073
- [Background] An Y, Wang G, Li X, Zhen Y, Zhao J, Li D. Rhinoplasty with Simultaneous Autologous Full-Face Fat Transfer for Asian Facial Contouring Balance: A Retrospective Study. Aesthetic Plast Surg. 2023 Apr;47(2):746-756. doi: 10.1007/s00266-022-03064-6. Epub 2022 Aug 30. PMID 36042025